CLINICAL TRIAL: NCT01280461
Title: An Open-label, Randomized, and Comparative Study to Evaluate the Efficacy and Safety of Cefoperazone/Sulbactam in Comparison to Cefepime for the Treatment of Hospital-acquired Pneumonia and Healthcare-associated Pneumonia
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Taipei Medical University WanFang Hospital (Other)
Responsible Party: Wen-Sen Lee, Department of Infectious Diseases, WanFang Hospital
Other Study IDs: 99067
Record Dates: First submitted 2011-01-19; First posted 2011-01-20 (Estimated); Last update posted 2011-01-20 (Estimated); Status verified 2011-01

CONDITIONS: Pneumonia
Keywords: Pneumonia
MeSH Terms: conditions — Pneumonia

STUDY DESIGN:
Observational Model: Cohort
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Experimental Group
- Control Group

SUMMARY:
This is a phase III, multi-center, open-label, comparative and randomized study in evaluating the efficacy and safety of cefoperazone/sulbactam versus cefepime for the treatment of hospital-acquired pneumonia and healthcare-associated pneumonia. The investigator will determine the total duration of study therapy, as clinically indicated. The minimum duration of study therapy will be 7 days and the maximum allowable duration of study therapy will be 21 days.

DETAILED DESCRIPTION:
Patients fulfill inclusion/exclusion criteria will be randomly assigned (in a 1:1 ratio)to receive intravenous cefoperazone/sulbactam or intravenous cefepime for 7~21days. Vitamin K1 10mg will be administered to cefoperazone/sulbactam group every 24 hours.

The assessment of clinical sign and symptoms of pneumonia and microbiological tests will be performed at early post-therapy visit and test-of-cure visit.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients aged ≧18 years old
* Patients with nosocomial bacterial pneumonia at least 48 hours after hospitalization or patients with healthcare-associated pneumonia(HCAP*).
* Clinical findings

At least two of the following signs:

1. Cough
2. Fever: axillary temperature > 37.5℃ or tympanic temperature > 38.5℃
3. Hypothermia: axillary temperature < 34℃ or tympanic temperature < 35℃
4. Purulent sputum production or respiratory secretion
5. Total peripheral white blood cell (WBC) count > 10,000/mm3; or > 15% band forms, regardless of total peripheral white count; or leucopenia with total WBC < 4500/mm3
6. Auscultatory findings on pulmonary examination of rales and/or evidence of pulmonary consolidation (dullness on percussion, bronchial breath sounds, or egophony)
7. Hypoxemia (defined as a partial O2 pressure <60 mmHg while the patient was breathing normal air or a decrease in the partial O2 pressure of ≧25% from an initial value)

   * Radiographic findings The chest radiograph should show the presence of a new or progressive infiltration on the chest X-ray film
   * Microbiologic criteria If sputum specimen is available and collected, both tests are mandatory with at least one of the following results is positive:

(1) Within 24 hours prior to, or at the time of enrollment, all patients should have had a culture and susceptibility testing of respiratory secretions or sputum to study drugs (2)Gram stain of respiratory secretions or sputum

* Patient must be able to sign a written informed consent form prior to the start of the study procedures. If any patient is unable to give consent, it must be obtained from the patient's legal representative
* Subject has not received more than 24 hours of a parenteral antibacterial drug for the current pneumonia. If subject has received more than 24 hours of a parenteral antibacterial drug, he/she must be declared as treatment failure.

Exclusion Criteria:

* Woman who are pregnant (determined by urine test) or lactating state
* Patients with known bronchial obstruction or a history of postobstructive pneumonia. (This does not exclude patients who have chronic obstructive pulmonary disease)
* A neutrophil count <1000/mm3
* Patients with pneumonia due to viral, fungal, or mycobacterial infection.
* Patients who were known to have been infected with human immunodeficiency virus
* Documented Legionella pneumonia
* Patients were infected with gram negative (G-) microorganism known to be resistant to one of the study antibiotics during trial
* Subjects with sputum gram stain of PMN>25, epithelial cell <10, and gram positive (G+) cocci in cluster predominant and phagocytosis
* Patients who have received any other investigational drug within 30 days prior to enrollment
* Patients who have received medications like cefoperazone, cefoperazone/sulbactam and cefepime within 30 days prior to enrollment
* Patients with abnormal pre-therapy laboratory data: aspartate aminotransferase (AST), alanine aminotransferase (ALT) ≧ 3X ULN (upper limit of normal); or serum creatinine, urea nitrogen > 3X ULN
* A history of hypersensitivity to penicillins, cephalosporins, carbapenems or J-lactam/J-lactamase inhibitors
* Severe disease (eg. septic shock, acute respiratory distress syndrome, and multiple organ failure) which may limit survival during therapy and follow-up period, or confound the results of the study as judged by the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with nosocomial bacterial pneumonia or healthcare-associated pneumonia(HCAP)
Sampling Method: Probability Sample
Enrollment: 142 (Estimated)
Dates: Start 2010-07; Study Completion 2011-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Wen-Sen Lee, Principal Investigator — Taipei Medical University WanFang Hospital
Locations (1):
- Taipei Medical University - WanFang Hospital, Taipei, Taiwan